CLINICAL TRIAL: NCT05720546
Title: Young Adult Infusion Space Survey: Comparing Experiences of Adolescents and Young Adults in Infusion Spaces at North Carolina Basnight Cancer Hospital
Brief Title: Young Adult Infusion Space Experience Satisfaction Survey
Status: Recruiting | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC2228
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Cancer
Keywords: Adolescent; survey
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Outpatient treatment center: Subjects received an infusion in an outpatient infusion center.
  Interventions: Other: Baseline Survey; Other: Semi-structured interviews; Other: Follow-up Survey
- Inpatient Infusion Center: Subjects received an infusion in an inpatient infusion center.
  Interventions: Other: Baseline Survey; Other: Semi-structured interviews; Other: Follow-up Survey

INTERVENTIONS:
Other: Baseline Survey — A survey that measures participant satisfaction will be offered to participants during infusion at baseline.
Other: Semi-structured interviews — Semi-structured interviews will be conducted in the same infusion spaces.
Other: Follow-up Survey — A survey that measures participant satisfaction will be offered to participants during following infusion.

SUMMARY:
The purpose of this study is to compare the satisfaction of Adolescent and Young Adults (AYA) receiving treatment in two different infusion spaces at the North Carolina Basnight Cancer Hospital (NCBCH). A survey and semi-structured interviews will be administered to participants to compare the experience with the built environment, with mental health staff, and between outpatient infusion spaces at NCBCH.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained to participate in the study and HIPAA authorization for the release of personal health information.
2. Subjects are willing and able to comply with study procedures based on the judgment of the investigator or protocol designee.
3. Age 18-39 years old at enrollment.
4. Receiving treatment for a cancer diagnosis in Adult Infusion Center or the Adolescent and Young Adult Infusion Center
5. English speaking.

Exclusion Criteria:

1. Dementia, altered mental status, or any psychiatric condition as determined by the clinical or study team that would prohibit the understanding or rendering of informed consent.
2. Current incarceration.

Ages: 18 Years to 39 Years | Sex: All
Age Groups: Adult
Study Population: A subject with a cancer diagnosis and receiving infusion in the study site
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
General satisfaction | Baseline (up to 1 month)
  General satisfaction will be measured with participants' responses to satisfaction surveys that will be administered in specific infusion spaces.
  Responses are rated on a Likert scale from 0 to 4. Scores will be summarized using frequency tables and percentages.

SECONDARY OUTCOMES:
Satisfaction with the built environment | Baseline (up to 1 month)
  Subject satisfaction with the built environment will be measured with a survey item specific to the built environment administered in specific infusion spaces. The result of satisfaction in different infusion sites will be compared.
  Responses are rated on a Likert scale from 0 to 2. Scores will be summarized using frequency tables and percentages.
Satisfaction with staff interaction | Baseline (up to 1 month)
  Subject satisfaction with staff interaction will be measured with a survey item specific to staff interactions administered in specific infusion spaces. The result of satisfaction in different infusion sites will be compared.
  Responses are rated on a Likert scale from 0 to 4. Scores will be summarized using frequency tables and percentages.
Satisfaction with mental health | Baseline (up to 1 month)
  Subject satisfaction with mental health will be measured with survey items regarding emotional support and comfort administered in specific infusion spaces. The result of satisfaction in different infusion sites will be compared.
  Responses are rated on a Likert scale from 0 to 4. Scores will be summarized using frequency tables and percentages.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Stein, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials